CLINICAL TRIAL: NCT01977131
Title: Phase 1 Study of Autologous Bone Marrow Stromal Cells With Modification by Hepatocyte Growth Factor to Treat Silicosis
Brief Title: Safety Study of Autologous Bone Marrow Stromal Cells With Modification by Hepatocyte Growth Factor to Treat Silicosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wei Yu (Other)
Responsible Party: Sponsor-Investigator, Wei Yu, Doctor, Guangzhou Municipal Twelfth People's Hospital
Organization: Guangzhou Municipal Twelfth People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010B031600019
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Silicosis
MeSH Terms: conditions — Silicosis | interventions — Cell Count

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stromal cells modified HGF (Experimental)
  Interventions: Other: Cells

INTERVENTIONS:
Other: Cells

SUMMARY:
The aim of this study was to analyze the safety, pulmonary function, and imaging changes of patients with silicosis treated with autologous bone marrow stromal cells with modification by hepatocyte growth factor.

ELIGIBILITY:
Inclusion Criteria:

- age between 18-50, chronic and accelerated silicosis, characterized with a fibrotic increase in the last two years, FEV1 <60% and > 40%, FVC > 60% and SaO2 >90%

Exclusion Criteria:

- smoking, active tuberculosis or other infections, cancer, auto-immune disorders, hematological, hepatic or cardiac diseases, and pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Absence of lung deficits during the procedure and/or in the 6 months follow-up | 6 months

SECONDARY OUTCOMES:
Improvement of pulmonary deficits | 1 year

REFERENCES:
- [Derived] Liu WW, Wang HX, Yu W, Bi XY, Chen JY, Chen LZ, Ding L, Han DM, Guo ZK, Lei YX. Treatment of silicosis with hepatocyte growth factor-modified autologous bone marrow stromal cells: a non-randomized study with follow-up. Genet Mol Res. 2015 Sep 9;14(3):10672-81. doi: 10.4238/2015.September.9.7. PMID 26400297